CLINICAL TRIAL: NCT07356193
Title: Effects of Lower Body Plyometric Training on Serum Creatine Phosphokinase and Creatinine Levels in Male Collegiate Volleyball Players
Brief Title: Serum CPK and Creatinine Changes During Plyometric Training in Collegiate Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Batterjee Medical College (Other)
Responsible Party: Principal Investigator, Mohamed A. Abdel Ghafar, Professor, Batterjee Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BMC-CPK-Study-2023
Record Dates: First submitted 2026-01-11; First posted 2026-01-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Muscle Damage; Plyometric Exercises; Creatine Kinase; Exercise Physiology
Keywords: Plyometric Training; Volleyball Players; Creatine Phosphokinase; Serum Creatinine
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lower Body Plyometric Training (Experimental)
  Interventions: Behavioral: Lower Body Plyometric Training; Other: control group
- Control Group (Active Comparator)
  Interventions: Other: control group

INTERVENTIONS:
Behavioral: Lower Body Plyometric Training — Training twice weekly for eight weeks, including low-, moderate-, and high-intensity plyometric exercises (squat jumps, box jumps, tuck jumps, split squat jumps, lateral hurdle jumps, zigzag jumps, single-leg tuck jumps, and depth jumps).
  Arms: Lower Body Plyometric Training
Other: control group — Routine volleyball training only; no plyometric exercises.

SUMMARY:
This retrospective study evaluated the effects of an eight-week lower body plyometric training program on serum creatine phosphokinase (CPK) and creatinine levels in male collegiate volleyball players. Sixty two players were divided into experimental and control groups. CPK and creatinine were measured at baseline and multiple time points during training. The study assessed whether plyometric training produced harmful biochemical changes or signs of rhabdomyolysis.

DETAILED DESCRIPTION:
This study evaluated the physiological effects and safety of an eight-week lower body plyometric training program in male collegiate volleyball players, focusing on changes in serum creatine phosphokinase (CPK) and creatinine levels. Sixty two healthy athletes were randomly assigned to either a plyometric training group or a control group. The experimental group performed progressive lower body plyometric exercises twice weekly for eight weeks, while the control group continued regular volleyball training.

Serum CPK and creatinine were assessed at baseline and multiple time points throughout the intervention. CPK levels in the training group increased significantly early in the program, peaking on Day 4 and remaining elevated until Week 2, before returning to baseline by Week 8. Importantly, all values remained within normal clinical ranges, and no signs of rhabdomyolysis or overtraining were observed. Serum creatinine levels showed no significant changes, indicating preserved renal function. No biomarker changes were detected in the control group.

These findings indicate that an eight-week, progressively designed plyometric training program is safe and well tolerated in male collegiate volleyball players.

ELIGIBILITY:
Inclusion Criteria:

* male collegiate volleyball players
* Age: 18-20 years
* No prior plyometric training

Exclusion Criteria:

* History of kidney disease
* Current musculoskeletal injury
* neuromuscular impairments

Ages: 18 Years to 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2022-02-13 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
Serum Creatine Phosphokinase (CPK) Levels | Baseline; Day 2; Day 4; Week 1; Week 2; Week 4; Week 6; Week 8
  Change in serum CPK measured using the CK-NAC optimized IFCC method.

SECONDARY OUTCOMES:
Serum Creatinine Levels | Baseline; Day 2; Day 4; Week 1; Week 2; Week 4; Week 6; Week 8
  Measured using modified Jaffe's method.

CONTACTS AND LOCATIONS:
Locations (1):
- Batterjee Medical College, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared because participant consent did not include permission for data sharing and the dataset contains sensitive physiological information.